CLINICAL TRIAL: NCT00667992
Title: A Phase 3, Randomised, Open-label, Crossover Study to Compare HFA vs CFC pMDI Formulations of Budesonide on Methacholine Hyper-reactivity in Patients With Stable, Persistent, Mild to Moderate Asthma
Brief Title: Study Comparing Budesonide Hydrofluoroalkane (HFA) vs Chlorofluorocarbon (CFC) Pressurized Metered Dose Inhalers (pMDI) in Patients With Mild to Moderate Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5252C00008
Record Dates: First submitted 2008-04-23; First posted 2008-04-28 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Asthma hyperreactivity
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide Hydrofluoroalkane (HFA) 100 (Active Comparator): Budesonide Hydrofluoroalkane (HFA) 100 mcg twice daily for 2 weeks
  Interventions: Drug: Budesonide HFA
- Budesonide HFA 400 (Active Comparator): Budesonide HFA 400 mcg twice daily for 2 weeks
  Interventions: Drug: Budesonide HFA
- Budesonide Chlorofluorocarbon (CFC) 100 (Active Comparator): Budesonide Chlorofluorocarbon(CFC) 100 mcg twice daily for 2 weeks
  Interventions: Drug: Budesonide CFC
- Budesonide CFC 400 (Active Comparator): Budesonide CFC 400 mcg twice daily for 2 weeks
  Interventions: Drug: Budesonide CFC

INTERVENTIONS:
Drug: Budesonide HFA — standard daily inhaled dose
  Arms: Budesonide HFA 400; Budesonide Hydrofluoroalkane (HFA) 100
Drug: Budesonide CFC — standard daily inhaled dose
  Arms: Budesonide CFC 400; Budesonide Chlorofluorocarbon (CFC) 100

SUMMARY:
This study is being carried out to see if budesonide with HFA is effective, safe and well tolerated compared with budesonide CFC. Budesonide HFA has been already given in other research studies, in both healthy volunteers and subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stable, persistent, mild to moderate asthma as defined by Global Initiative for Asthma (GINA) Guidelines and for whom FEV1 > 60 %
* ICS taking ≤ 1000 μg BDP per day, or equivalent
* Methacholine PC20 < 4 mg/mL

Exclusion Criteria:

* Known or suspected hypersensitivity to budesonide or any other constituents of the budesonide HFA pMDI or budesonide CFC pMDI.
* Currently a smoker or who has ceased smoking within 6 months of Visit 1.
* Exacerbations of asthma requiring oral steroids, hospitalisation or change in asthma therapy in the previous three months.
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or bronchiectasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, PhD, MD, Principal Investigator — Asthma and Allergy Research Group Division of Medicine and Therapeutics Ninewells Hospital and Medical School University of Dundee
Locations (3):
- Research Site, King of Prussia, Pennsylvania, United States
- United Kingdom (2):
  - Research Site, Dundee, Scotland
  - Research Site, Perth, Scotland

REFERENCES:
- [Derived] Anderson WJ, Short PM, Jabbal S, Lipworth BJ. Inhaled corticosteroid dose response in asthma: Should we measure inflammation? Ann Allergy Asthma Immunol. 2017 Feb;118(2):179-185. doi: 10.1016/j.anai.2016.11.018. Epub 2017 Jan 3. PMID 28065396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 144 were enrolled, 45 were excluded: 11 for eligibility not fulfilled, 8 with condition under investigation worsened, 8 for voluntary withdrawal, 17 with reasons not specified, and 1 lost to follow-up and 99 were randomised.
Groups:
- Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC: Budesonide Hydrofluoroalkane (HFA), 100 mcg twice daily followed by Budesonide HFA 400 mcg twice daily First, Wash out, then Budesonide Chlorofluorocarbon (CFC) 100 mcg twice daily followed by Budesonide CFC 400 mcg twice daily.
- Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA: Budesonide CFC, 100 mcg twice daily followed by Budesonide CFC 400 mcg twice daily First, Wash out, then Budesonide HFA 100 mcg twice daily followed by 400 mcg twice daily.
Period: First Intervention 100 Mcg Twice Daily
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA
Started | 49 | 50
Completed | 44 | 45
Not Completed | 5 | 5
Not completed — Condition Under Investigation Worsened | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervention 400 Mcg Twice Daily
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA
Started | 44 | 45
Completed | 41 | 41
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Condition Under Investigation Worsened | 2 | 3
Not completed — Medication not allowed taken | 0 | 1
Period: Wash-out
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA
Started | 41 | 41
Completed | 34 | 36
Not Completed | 7 | 5
Not completed — Not within one doubling dilution | 4 | 3
Not completed — Failure to wash-out | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Third Intervention 100 Mcg Twice Daily
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA
Started | 34 | 36
Completed | 33 | 35
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Forth Intervention 400 Mcg Twice Daily
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA
Started | 33 | 35
Completed | 33 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC: Budesonide Hydrofluoroalkane (HFA), 100 mcg twice daily followed by Budesonide HFA 400 mcg twice daily, First then Budesonide Chlorofluorocarbon (CFC) 100 mcg twice daily followed by Budesonide CFC 400 mcg twice daily.
- Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA: Budesonide CFC, 100 mcg twice daily followed by Budesonide CFC 400 mcg twice daily First, then Budesonide HFA 100 mcg twice daily followed by 400 mcg twice daily.
- Total: Total of all reporting groups
Arm/Group | Budesonide Hydrofluoroalkane (HFA) First, Then Budesonide CFC | Budesonide Chlorofluorocarbon (CFC) First, Then Budesonide HFA | Total
Number analyzed (Participants) | 44 | 45 | 89
Age Continuous [Mean (Full Range); unit: years] | 40.0 [19.0 to 65.0] | 39.5 [18.0 to 64.0] | 39.75 [18.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: PC 20 Methacholine (Provocative Concentration of Methacholine Causing 20 % Fall in FEV1(Forced Expiratory Volume)
Description: Provocative concentration of methacholine is that causing a 20% fall in FEV1. The methacholine challenge test entailed the patient inhaling from an aerosol containing doubling concentrations of methacholine over a period of 2 minutes until FEV1 had been reduced by 20%.
  The ratio of Methacholine concentration measured at 2 weeks to that at Baseline.
Time Frame: Baseline and week 2
Population: Full analysis set (FAS). The FAS was defined as all randomised patients who contributed data from at least one period (ie data from both low and high dose of one inhaler).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Budesonide Chlorofluorocarbon(CFC) 100: Budesonide Chlorofluorocarbon (CFC) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon(CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Ratio | 1.546 [1.343 to 1.780] | 2.163 [1.877 to 2.494] | 1.673 [1.449 to 1.928] | 2.079 [1.801 to 2.401]

2. Secondary Outcome: Peak Exploratory Flow (PEF)
Description: Change in PEF at Week 2 from baseline, mean over all days in run-in and all dasy in treatment period, with baseline as covariate.
Time Frame: Baseline to week 2 recorded daily
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minutes
Groups:
- Budesonide Chlorofluorocarbon(CFC) 100: Budesonide Chlorofluorocarbon(CFC) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon(CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Liters/minutes | 9.7 [3.9 to 15.6] | 12.7 [6.8 to 18.6] | 12.0 [6.1 to 17.9] | 9.1 [3.2 to 15.1]

3. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second)
Description: FEV1 change from baseline
Time Frame: Baseline to week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Budesonide Hydrofluoroalkane(HFA) 100: Budesonide Hydrofluoroalkane(HFA) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Liters | 0.08 [0.05 to 0.11] | 0.10 [0.07 to 0.13] | 0.10 [0.07 to 0.13] | 0.11 [0.08 to 0.14]

4. Secondary Outcome: FEF 25-75 (Forced Expiratory Flow 25-75)
Description: FEF 25-75- Forced expiratory flow over the middle one half of the FVC. The results are expressed as the change from baseline
Time Frame: Baseline and week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/seconds
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Liters/seconds | 0.11 [0.005 to 0.17] | 0.14 [0.08 to 0.20] | 0.15 [0.09 to 0.21] | 0.20 [0.13 to 0.26]

5. Secondary Outcome: eNO (Exhaled Nitrogen Oxide)
Description: eNO ratio of baseline
Time Frame: baseline and week 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Budesonide Chlorofluorocarbon (CFC) 100: Budesonide Chlorofluorocarbon (CFC) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Ratio | 0.66 [0.62 to 0.70] | 0.57 [0.53 to 0.60] | 0.66 [0.63 to 0.70] | 0.59 [0.55 to 0.62]

6. Secondary Outcome: Asthma Symptom Score Morning
Description: Asthma Symptom score recorded daily in the morning: Scale: 0-3. 0 = None; no asthma symptoms. 1 = Mild symptoms; aware of asthma symptoms but easily tolerated. 2 = Moderate symptoms; asthma causing enough discomfort to cause problems with normal activities (or with sleep). 3 =Severe symptoms; unable to do normal activities. The average of means for values recorded daily in the morning is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon(CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Units on a scale | 0.39 [0.34 to 0.44] | 0.29 [0.24 to 0.34] | 0.39 [0.34 to 0.44] | 0.30 [0.25 to 0.35]

7. Secondary Outcome: Asthma Symptom Score Evening
Description: Asthma Symptom score recorded daily in the evening: Scale: 0-3. 0 = None; no asthma symptoms. 1 = Mild symptoms; aware of asthma symptoms but easily tolerated. 2 = Moderate symptoms; asthma causing enough discomfort to cause problems with normal activities (or with sleep). 3 =Severe symptoms; unable to do normal activities. The average of means for values recorded daily in the evening is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Budesonide Hydrofluoroalkane(HFA) 100: Budesonide Hydrofluoroalkane (HFA) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Units on a scale | 0.48 [0.43 to 0.52] | 0.32 [0.27 to 0.38] | 0.46 [0.41 to 0.50] | 0.36 [0.31 to 0.41]

8. Secondary Outcome: Asthma Symptom Score Total
Description: Asthma Symptom score recoded daily, Total. Scale: 0 - 3. 0 = None; no asthma symptoms. 1 = Mild symptoms; aware of asthma symptoms but easily tolerated. 2 = Moderate symptoms; asthma causing enough discomfort to cause problems with normal activities (or with sleep). 3 =Severe symptoms; unable to do normal activities. The average of means for values recorded daily is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Units on a scale | 0.87 [0.78 to 0.96] | 0.61 [0.52 to 0.71] | 0.85 [0.76 to 0.94] | 0.66 [0.56 to 0.76]

9. Secondary Outcome: Rescue Medication Morning
Description: The average of means for inhalations of rescue medication in the morning is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations
Groups:
- Budesonide Hydrofluoroalkane (HFA) 100: Budesonide Hydrofluoroalkane(HFA) 100 mcg twice daily for 2 weeks
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Number of inhalations | 0.71 [0.60 to 0.82] | 0.45 [0.34 to 0.56] | 0.62 [0.51 to 0.73] | 0.50 [0.39 to 0.61]

10. Secondary Outcome: Rescue Medication Evening
Description: The average of means for inhalations of rescue medication in the evening is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations
Arm/Group | Budesonide Hydrofluoroalkane(HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Number of inhalations | 0.90 [0.77 to 1.03] | 0.67 [0.52 to 0.80] | 0.84 [0.71 to 0.97] | 0.64 [0.50 to 0.78]

11. Secondary Outcome: Rescue Medication Total
Description: The average of means for inhalations of rescue medication in morning and evening combined over a 24 hour period is presented.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations/24 hours
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon(CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Number of inhalations/24 hours | 1.58 [1.35 to 1.80] | 1.10 [0.86 to 1.33] | 1.39 [1.16 to 1.62] | 1.05 [0.81 to 1.29]

12. Secondary Outcome: Peak Exploratory Flow (PEF) Morning
Description: Peak Exploratory Flow (PEF) recorded daily in the morning
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minutes
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Number analyzed (Participants) | 80 | 79 | 79 | 78
Liters/minutes | 426 [421 to 431] | 437 [433 to 442] | 428 [424 to 433] | 438 [433 to 442]

ADVERSE EVENTS:
Arm/Group | Budesonide Hydrofluoroalkane (HFA) 100 | Budesonide HFA 400 | Budesonide Chlorofluorocarbon (CFC) 100 | Budesonide CFC 400
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/81 | 2/85 | 0/79
Other Adverse Events (participants affected / at risk) | 0/86 | 0/81 | 0/85 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide Hydrofluoroalkane (HFA) 100 (N=86) | Budesonide HFA 400 (N=81) | Budesonide Chlorofluorocarbon (CFC) 100 (N=85) | Budesonide CFC 400 (N=79)
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No